CLINICAL TRIAL: NCT01088958
Title: Diarrhea, Malaria, Anemia, and Helminthiasis Prevention Through Household-based Interventions in Rural Western Kenya: the Nyando Integrated Child Health and Education (NICHE) Project
Brief Title: Effectiveness of Selling Micronutrient Sprinkles in Rural Kenya
Acronym: NICHE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Safe Water and AIDS Project (Other); Kenya Medical Research Institute (Other); Global Alliance for Improved Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-5039
Record Dates: First submitted 2010-02-26; First posted 2010-03-18 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Anemia, Iron-deficiency
Keywords: Kenya; Child Nutrition Disorders; Social marketing
MeSH Terms: conditions — Anemia, Iron-Deficiency; Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micronutrient Sprinkles (Experimental): Sales of Sprinkles in these groups of villages by community vendors
  Interventions: Dietary Supplement: Micronutrient powders (Sprinkles)

INTERVENTIONS:
Dietary Supplement: Micronutrient powders (Sprinkles) — Sprinkles were developed in 1996 by Stanley Zlotkin's research group at the Hospital for Sick Children, University of Toronto as a novel approach for delivering iron and other micronutrients. They come in 1g sachets of dry powder that is then added to any home-prepared semi-solid food, intended for daily consumption by children aged 6-59 months. Formulation includes:
  Iron (Ferrous fumarate) 12.5 mg, Folic acid 150 µg, Vitamin A 375 µg, Vitamin C 35 mg, Zinc 5 mg, Vitamin B1 0.5 mg, Vitamin B2 0.5 mg, Vitamin B6 0.5 mg, Vitamin B12 0.9 µg, Vitamin D3 5 µg, Vitamin E 6.0 mg, Niacin 6.0 mg, Copper 0.6 mg, Iodine 50 µg

SUMMARY:
The purpose of the study is to evaluate the effectiveness of household-based distribution of evidence-based health products and to measure the health impact of these combined interventions on a population basis.

DETAILED DESCRIPTION:
Nyanza Province has the highest mortality rates for infants and children under 5 years of age and the highest HIV prevalence rates in Kenya. Burden of disease in western Kenya is further characterized by endemic malaria transmission, diarrheal diseases due to poor access to safe water, and iron deficiency anemia (IDA) in over 60% of children. Access to health interventions in rural Nyanza Province is poor due to limited transportation and communication infrastructure. Delivery of household-based interventions through local institutions offers the potential for increased utilization and improved health outcomes in rural areas. The Centers for Disease Control and Prevention (CDC) in partnership with the Rotary-supported Safe Water and AIDS Project (SWAP), initiated a program in 2007 that combines household, clinic, school, and local commercial distribution approaches to increase access to various evidence-based health products (WaterGuard(TM) and PuR(TM) water disinfectant products, water storage containers, soap, insecticide treated bednets, micronutrient Sprinkles(TM), and albendazole) and measures the health impact of these combined interventions on a population basis.

Evaluation of the intervention will take place over 36 months and will include: 1) baseline and follow-up cross sectional surveys among households in communities visited by SWAP for purchase of products; 2) active household surveillance of diarrhea, febrile illness and Sprinkles(TM) usage; 3) testing of hemoglobin and iron status and anthropometry measurement among children aged 6-35 months; 4) focus groups and targeted interviews to assess the acceptability of health products; and 5) other program evaluation methods.

During the baseline and follow-up surveys, demographic information, water, sanitation, hygiene, and health information, dietary intake history, and other data will be collected by questionnaire. A blood specimen collected by fingerstick will be used to test for hemoglobin concentration, malaria parasitemia, and iron status. Follow-up surveys 12 and 24 months after baseline data collection will include collection of similar data to assess the effectiveness of product distribution. Anthropometry will be measured at baseline, 12, and 24 months. Qualitative information on user preferences will be obtained using ongoing focus groups, observations and targeted interviews. The results of these evaluations will be published in reports distributed to SWAP, the Kenyan government, and local NGO's and in peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-36 months at the time of enrollment
* Live within the study area for the duration of the intervention and follow-up period

Exclusion Criteria:

* Unavailable for enrollment on 3 separate household visits
* Parental refusal to give informed consent

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7200 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Product sales and use (coverage) | Every 2 weeks
  Biweekly household visits of selected cohort take place to assess purchases and use of health products and self reported morbidity outcomes. Household visits started at enrollment and continued throughout 2-year study period.

SECONDARY OUTCOMES:
Prevalence of anemia | Baseline and 12 and 24-month follow-up surveys
Prevalence of iron deficiency | Baseline and 12 and 24-month follow-up surveys

CONTACTS AND LOCATIONS:
Overall Officials: Parminder S Suchdev, MD MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC/Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Result] Centers for Disease Control and Prevention (CDC). Baseline data from the Nyando Integrated Child Health and Education Project--Kenya, 2007. MMWR Morb Mortal Wkly Rep. 2007 Oct 26;56(42):1109-13. PMID 17962803
- [Result] Suchdev PS, Leeds IL, McFarland DA, Flores R. Is it time to change guidelines for iron supplementation in malarial areas? J Nutr. 2010 Apr;140(4):875-6. doi: 10.3945/jn.109.118638. Epub 2010 Feb 10. No abstract available. PMID 20147465
- [Result] Suchdev PS, Ruth L, Obure A, Were V, Ochieng C, Ogange L, Owuor M, Ngure F, Quick R, Juliao P, Jung C, Teates K, Cruz K, Jefferds ME. Monitoring the marketing, distribution, and use of Sprinkles micronutrient powders in rural western Kenya. Food Nutr Bull. 2010 Jun;31(2 Suppl):S168-78. doi: 10.1177/15648265100312S209. PMID 20715601
- [Derived] Davis JN, Williams A, Arnold CD, Rohner F, Wirth JP, Addo Y, Flores-Ayala RC, Oaks BM, Young MF, Suchdev PS, Engle-Stone R. The Relationship Between Ferritin and BMI is Mediated by Inflammation Among Women in Higher-Income Countries, But Not in Most Lower-Income Countries Nor Among Young Children: A Multi-Country Analysis. Curr Dev Nutr. 2022 Sep 9;6(10):nzac139. doi: 10.1093/cdn/nzac139. eCollection 2022 Oct. PMID 36475018
- [Derived] Suchdev PS, Addo OY, Martorell R, Grant FK, Ruth LJ, Patel MK, Juliao PC, Quick R, Flores-Ayala R. Effects of community-based sales of micronutrient powders on morbidity episodes in preschool children in Western Kenya. Am J Clin Nutr. 2016 Mar;103(3):934-41. doi: 10.3945/ajcn.115.118000. Epub 2016 Feb 10. PMID 26864367
- [Derived] Suchdev PS, Ruth LJ, Woodruff BA, Mbakaya C, Mandava U, Flores-Ayala R, Jefferds ME, Quick R. Selling Sprinkles micronutrient powder reduces anemia, iron deficiency, and vitamin A deficiency in young children in Western Kenya: a cluster-randomized controlled trial. Am J Clin Nutr. 2012 May;95(5):1223-30. doi: 10.3945/ajcn.111.030072. Epub 2012 Apr 4. PMID 22492366
- [Derived] Grant FK, Martorell R, Flores-Ayala R, Cole CR, Ruth LJ, Ramakrishnan U, Suchdev PS. Comparison of indicators of iron deficiency in Kenyan children. Am J Clin Nutr. 2012 May;95(5):1231-7. doi: 10.3945/ajcn.111.029900. Epub 2012 Mar 28. PMID 22456661
- See also: Implementing NGO — http://www.swapkenya.org/